CLINICAL TRIAL: NCT04485728
Title: Sleep Improvement Intervention for Hospitalized Antepartum Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sam Houston State University (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other); Memorial Hermann Texas Medical Center (Unknown)
Responsible Party: Principal Investigator, Andrea Smith, Assistant Professor, Sam Houston State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2020-83
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Sleep Disturbance in Hospitalized Antepartum Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Improvement Intervention (Experimental)
  Interventions: Behavioral: Sleep Improvement Protocol Intervention for Hospitalized Antepartum Patients
- Standard of Care (Control) (No Intervention)

INTERVENTIONS:
Behavioral: Sleep Improvement Protocol Intervention for Hospitalized Antepartum Patients — Patients are getting sleep hygiene education and a sleep hygiene kit.
  Arms: Sleep Improvement Intervention

SUMMARY:
This project seeks to further study the effects of a hospital-based protocol for improving sleep in high-risk antepartum patients as piloted by Lee and Gay (2017).

ELIGIBILITY:
Inclusion Criteria:

* speak, read, and write English
* medically stable
* 20 weeks' gestation or greater
* viable fetus
* hospitalized at least 24 hours

Exclusion Criteria:

* Do not speak, read, and write English
* Medically unstable
* Less than 20 weeks' gestation
* Nonviable fetus
* Hospitalized less than 24 hours

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Number of patients who use the sleep improvement intervention | Day 7
Level of satisfaction with the intervention as assessed by a Likert assessment | Day 7
  The scale ranges from 0-5 with 5 being extremely satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Smith, Ph.D., RN, Principal Investigator — Sam Houston State University
Locations (1):
- Memorial Hermann Texas Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No